CLINICAL TRIAL: NCT00999804
Title: TBCRC 023: A Randomized Multicenter Phase II Neoadjuvant Trial of Lapatinib Pus Trastuzumab, With or Without Endocrine Therapy for 12 Weeks vs. 24 Weeks in Patients With HER2 Overexpressing Breast Cancer
Brief Title: Extension Study of Lapatinib Plus Herceptin With or Without Endocrine Therapy
Acronym: HELEX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Professor, Baylor Breast Care Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25846
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Locally Advanced Breast Cancer Neoadjuvant Endocrine
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Letrozole; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24-week arm (Experimental): Participants will receive 24-weeks of lapatinib plus trastuzumab. Participants who are estrogen receptor (ER) and/or progesterone receptor (PR) positive will also receive endocrine therapy.
  Interventions: Drug: Lapatinib; Drug: Letrozole; Drug: Trastuzumab
- 12-week arm (Active Comparator): Participants will receive 12-weeks of lapatinib plus trastuzumab. Participants who are estrogen receptor (ER) and/or progesterone receptor (PR) positive will also receive endocrine therapy.
  Interventions: Drug: Lapatinib; Drug: Letrozole; Drug: Trastuzumab

INTERVENTIONS:
Drug: Lapatinib — 1000 mg of Lapatinib by mouth daily
  Other Names: TyKerb
Drug: Letrozole — Letrozole, 2.5 mg by mouth daily (for hormone receptor positive participants only)
  Other Names: Femara
Drug: Trastuzumab — 6 mg/kg intravenously, every 3 weeks
  Other Names: Herceptin

SUMMARY:
Breast cancer is the most common malignancy in the U.S. Targeted therapies such as tamoxifen have been revolutionary in reducing tumor recurrences and mortality in early breast cancer. Using this successful paradigm, there has been a continued search for other targeted biologic therapies directed at receptors with known potential for promoting tumor growth.

The estrogen receptor (ER) and/or the HER signaling pathways are the dominant drivers of cell proliferation and survival in the majority of human breast cancers. Molecular targets of these pathways provide the most effective therapies in appropriately selected patients. However, de novo and acquired resistance remain major obstacles to successful treatment, and understanding the molecular pathways responsible for this resistance would enable the discovery of new strategies to overcome it.

The superiority of multi-drug HER2-targeted therapy over single agent therapy has been demonstrated in the preclinical setting using mouse xenografts. Trastuzumab, pertuzumab, lapatinib, and gefitinib, represent a group of therapeutic agents that target the HER family by different molecular mechanisms. Used as single agents in the MCF7/HER2-18 xenograft model, these drugs restored or enhanced sensitivity to tamoxifen. However, tumor growth inhibition lasted only 2-3 months before resistance to treatments occurred. However, when gefitinib, a HER1 inhibitor, was added to the two-antibody (T+P) regimen to block signals from HER1 dimers, a complete disappearance of nearly all xenograft tumors was observed; moreover, there was evidence of complete tumor eradication in 50% of the mice. The combination of lapatinib + trastuzumab was also highly effective in eradication of tumor burden, with no evidence of re-growth after 200 days. These xenograft models demonstrate that multi-drug HER2-targeted therapy more effectively induces apoptosis and inhibits proliferation, thereby resulting in tumor regression. Furthermore, HER2 combination therapy appears to more effectively reduce levels of phosphorylated pAKT and MAPK, thus resulting in sustained tumor inhibition.

DETAILED DESCRIPTION:
Breast cancer cells have certain characteristics or traits--these traits are called biomarkers. There are three biomarkers that help doctors decide which treatment to give any given patient. These biomarkers are the estrogen receptor (ER), progesterone receptor (PgR), and HER2 protein. Breast cancer cells that have a large number of estrogen or progesterone receptors are called ER and/or PgR positive. Cancers that are ER and/or PgR positive use the hormones estrogen and progesterone to help them grow. Not all breast cancers are ER or PgR positive. Patients are being asked to take part in this study that have a special type of breast cancer called HER2 positive breast cancer. HER2-positive breast cancer is a breast cancer that tests positive for a protein called human epidermal growth factor receptor-2 (HER2). HER2 is located on the outer surface of a cancer cell. The HER2 protein sends a signal to the inside of the cancer cells telling it to grow and divide.

Two medications that directly target this HER2 protein. One is called trastuzumab(Herceptin), and the other is called lapatinib (Tykerb). Both medications are FDA-approved for the treatment of women with HER2+ breast cancer. Each medication attaches to the protein so that it can no longer function. Once the protein stops working, the cancer cells can no longer make copies of themselves. This makes cancer shrink. Both drugs target HER2; however each drug works a little bit differently.

Some patients respond better to Herceptin, and some patients respond better to Tykerb. Right now, we are not sure why some patients respond to one drug but do not respond to the other drug. One possibility is that in some patients, the HER2 protein finds another way to send its message to the inside of the cell (similar to a road detour). For example, when one path is "closed" because the drug is blocking it, the HER2 protein finds a different way to send its signal. We think that we can completely block the HER2 protein by giving patients both Tykerb and Herceptin.

Some patients with HER positive breast cancer are also ER and/or PgR positive. Even after HER2 is completely blocked, these types of cancer cells can still grow by using the estrogen or progesterone receptor. If a patient is told they are ER and/or PgR positive, they will also take an anti-estrogen pill along with Tykerb and Herceptin. We think that we can stop cancer growth more completely by blocking both the HER2 protein and the ER/PR receptors.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female and at least 18 years of age.
2. Signed informed consent.
3. Locally advanced breast cancers are eligible. Locally advanced cancers must be of clinical and/or radiologic size >3 cm, or >2 cm with clinical evidence of axillary nodal involvement*. (If tumors are less than 3 cm, we will use the radiologically measured tumor size to determine if the tumor meets the minimal size requirements.)
4. Patients must have histologically confirmed invasive mammary carcinoma that is HER2 overexpressing, defined as 3+ by immunohistochemistry, or a FISH/CEP ratio greater than 2.
5. Negative serum pregnancy test (HCG) within 7 days of starting study drug, if of child-bearing potential.
6. Kidney and liver function tests - all within 1.5 times the institutional upper limit of normal.
7. Performance status (WHO/ECOG scale) 0-1 and life expectancy >6 months.
8. No evidence of brain or leptomeningeal disease, or any other Stage IV disease.
9. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

1. Patients with bilateral breast cancer.
2. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
3. Severe underlying chronic illness or disease.
4. Cardiomyopathy or baseline LVEF less than 50%.
5. Other investigational drugs while on study.
6. Severe or uncontrolled hypertension, history of congestive heart failure or severe coronary arterial disease.
7. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded
8. Taking any lapatinib prohibited medication(s)
9. Inability or unwillingness to comply with, or follow study procedures.
10. Patients who have received any form of treatment for breast cancer within the past five years, including surgical resection, chemotherapy, endocrine therapy, or biologic therapy.
11. Patients with a prior history of ipsilateral invasive breast cancer or carcinoma in situ who present with a new primary.
12. Patients with known active, infectious Hepatitis B, Hepatitis C, or HIV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (8):
- United States (8):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine Lester and Sue Smith Breast Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rimawi MF, Niravath P, Wang T, Rexer BN, Forero A, Wolff AC, Nanda R, Storniolo AM, Krop I, Goetz MP, Nangia JR, Jiralerspong S, Pavlick A, Veeraraghavan J, De Angelis C, Gutierrez C, Schiff R, Hilsenbeck SG, Osborne CK; Translational Breast Cancer Research Consortium. TBCRC023: A Randomized Phase II Neoadjuvant Trial of Lapatinib Plus Trastuzumab Without Chemotherapy for 12 versus 24 Weeks in Patients with HER2-Positive Breast Cancer. Clin Cancer Res. 2020 Feb 15;26(4):821-827. doi: 10.1158/1078-0432.CCR-19-0851. Epub 2019 Oct 29. PMID 31662331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between October 2011 and July 2014 at 10 study sites: Baylor College of Medicine, UAB, University of Chicago, Johns Hopkins, Duke, Indiana University, Vanderbilt, MDACC, DFCI, and Mayo Clinic.
Pre-assignment Details: Participants screened up to 28-day period.
Groups:
- 24-week Arm: Participants will receive 24-weeks of lapatinib plus trastuzumab. Participants who are estrogen receptor (ER) and/or progesterone receptor (PR) positive will also receive endocrine therapy.
  Lapatinib: 1000 mg by mouth daily
  Letrozole: 2.5 mg by mouth daily (for hormone receptor positive participants only)
  Trastuzumab: 6 mg/kg intravenously, every 3 weeks
- 12-week Arm: Participants will receive 12-weeks of lapatinib plus trastuzumab. Participants who are estrogen receptor (ER) and/or progesterone receptor (PR) positive will also receive endocrine therapy.
  Lapatinib: 1000 mg by mouth daily
  Letrozole: 2.5 mg by mouth daily (for hormone receptor positive participants only)
  Trastuzumab: 6 mg/kg intravenously, every 3 weeks
Period: Overall Study
Arm/Group | 24-week Arm | 12-week Arm
Started | 85 | 43
Completed | 64 | 38
Not Completed | 21 | 5
Not completed — Lack of Efficacy | 9 | 2
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Death | 1 | 0
Not completed — Ineligible | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-week Arm | 12-week Arm | Total
Number analyzed (Participants) | 85 | 43 | 128
Age, Continuous [Median (Full Range); unit: years] | 50 [23 to 80] | 57 [38 to 88] | 52 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 43 | 128
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 69 | 33 | 102
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 10 | 21
  White | 68 | 31 | 99
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: Pathologic complete response was defined as no residual invasive cancer in the breast, after 12 or 24 weeks of lapatinib/trastuzumab with or without endocrine therapy.
  This outcome is based on patient's pathological report. We are not measuring the clinical response.
  Participants who have received at least one cycle of therapy (defined as one dose of trastuzumab and 21 days of lapatinib), and have had their response classified were evaluable.
Time Frame: 12 or 24 week depending the arm assignment
Population: Participants who have received at least one cycle of therapy (defined as one dose of trastuzumab and 21 days of lapatinib), and have had their response classified were evaluable. 4 participant were not evaluable: 3 participant were found ineligible for the study and one participant died before surgery.
Measure: Number; unit: participants
Arm/Group | 24-week Arm | 12-week Arm
Number analyzed (Participants) | 81 | 43
participants
  pathologic complete response | 20 | 5
  non-complete pathologic response | 61 | 38
Statistical Analysis 1: Comparison: 24-week Arm; The study was planned to enroll 136 patients if the original cohort (n=90) was deemed successful. The 24 weeks arm ran as a single arm, using an admissible Simon-like two-stage design. The 12 weeks arm accrued as long as the 24 weeks arm is open. The analysis of the first cohort indicated that 15 pCR were observed , which did not meet the required 20 or more responses. The accrual was closed early and the study has a total of 128 participants; Test type: Superiority or Other; proportion of pCR = 0.25 — No comparison is required between the 24 weeks arm and 12 weeks arm. The study is designed as the 24 weeks arm ran as a single arm, using an admissible Simon-like two-stage design and required 20 or more responses in the first 55 evaluable patients

2. Secondary Outcome: Number of Participants With Adverse Events
Description: the safety and tolerability of an extended regimen of lapatinib + trastuzumab, with or without endocrine therapy
Time Frame: 12 week or 24 weeks depending on arm assignment
Population: Participants who started the study treatment will be evaluable for safety analysis
Measure: Number; unit: participants
Arm/Group | 24-week Arm | 12-week Arm
Number analyzed (Participants) | 85 | 43
participants | 61 | 26
Statistical Analysis 1: Comparison: 24-week Arm; This outcome is to establish the safety and tolerability of an extended regimen of lapatinib + trastuzumab, with or without endocrine therapy. No comparison between the 2 arms is required; Test type: Superiority or Other; proportion of patients with AE = 0.72 — 61 out of 85 patients (72%) in the 24-week arm had at least 1 adverse events

3. Secondary Outcome: Total Pathologic Complete Response
Description: pathologic complete response was defined as no residual invasive cancer in the breast and the axillary lymph nodes.
Time Frame: 12 weeks or 24 weeks depending on arm assignment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 24-week Arm | 12-week Arm
Number analyzed (Participants) | 81 | 43
participants
  total complete pathologic response | 8 | 2
  not total complete pathologic response | 72 | 41
Statistical Analysis 1: Comparison: 24-week Arm; No comparison between the two arms is required; Test type: Superiority or Other; proportion of tpCR in 24 weeks arm = 0.1

4. Secondary Outcome: Clinical Response
Time Frame: 12 weeks or 24 weeks depending on arm assignment
Population: Participants who have received at least one cycle of therapy (defined as one dose of trastuzumab and 21 days of lapatinib), and have had their response classified were evaluable. 4 participants were not evaluable for efficacy.
Measure: Number; unit: participants
Arm/Group | 24-week Arm | 12-week Arm
Number analyzed (Participants) | 81 | 43
participants
  Complete response | 46 | 21
  Partial response | 10 | 13
  Stable disease | 2 | 3
  Progressive disease | 13 | 4
  Unknown | 10 | 2
Statistical Analysis 1: Comparison: 24-week Arm; No comparison between the 2 arm is required for this study; Test type: Superiority or Other; proportion of CR+PR in 24 weeks arm = 0.69

ADVERSE EVENTS:
Time Frame: 7 months
Description: Adverse events experienced by participants will be collected and reported from initiation of study medication, throughout the study, and within 30 days of the last dose of study medication.
Arm/Group | 24-week Arm | 12-week Arm
Serious Adverse Events (participants affected / at risk) | 3/85 | 1/43
Other Adverse Events (participants affected / at risk) | 61/85 | 26/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-week Arm (N=85) | 12-week Arm (N=43)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Elevated AST (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-week Arm (N=85) | 12-week Arm (N=43)
Alanine aminotransferase increased (Investigations) | 22 (54) | 5 (7)
Alkaline phosphatase increased (Investigations) | 12 (17) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 8 (16) | 4 (11)
Anorexia (Metabolism and nutrition disorders) | 8 (10) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 23 (46) | 7 (7)
Blood bilirubin increased (Investigations) | 8 (15) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 30 (51) | 14 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 14 (19) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Hot flashes (Vascular disorders) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 9 (15) | 10 (10)
Nusea (General disorders) | 11 (15) | 6 (6)
Pain (General disorders) | 5 (6) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 17 (22) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (11) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No